CLINICAL TRIAL: NCT05378516
Title: Placental Pathology and Inflammatory Factor Analysis of Obstetric Antiphospholipid Syndrome Patients
Brief Title: Placental Pathology and Inflammatory Factor Analysis of OAPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yang Jingjing, Deputy chief physician, Peking University People's Hospital
Other Study IDs: yjjbear2022
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-01

CONDITIONS: Antiphospholipid Syndrome in Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- obstetric antiphospholipid syndrome: obstetric antiphospholipid syndrome 20 cases and normal pregnant women 20 cases
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This investigation is on placental pathological changes and inflammatory factors associated with obstetric antiphospholipid syndrome.

DETAILED DESCRIPTION:
1. To clarify the correlation between antiphospholipid antibody, ACC1 expression level, Treg cell and placental pathological changes associated with antiphospholipid syndrome. 2. Reveal that antiphospholipid antibodies affect Treg cell differentiation through the key enzyme of lipid metabolism ACC1.

ELIGIBILITY:
Inclusion Criteria:

1. pregnant women with antiphospholipid syndrome (diagnosed by experts with clinical evidence) and healthy pregnant women without antiphospholipid syndrome as a control group
2. consent to join this study and finish the informed consents

Exclusion Criteria:

pregnant women with other autoimmune diseases

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women with antiphospholipid syndrome (diagnosed by experts with clinical evidence) and healthy pregnant women without antiphospholipid syndrome as a control group
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
expression of ACC1 in placenta in pregnancy with/without antiphospholipid syndrome | in two years

CONTACTS AND LOCATIONS:
Overall Officials: Jingjing Yang, doctor, Principal Investigator — Peking University People's Hospital
Locations (1):
- PekingUPH, Beijing, China

IPD SHARING:
Plan to Share IPD: No